CLINICAL TRIAL: NCT05333302
Title: Pilot Study of CD19 CAR-T Cells Therapy for Relapsed or Refractory Acute Lymphoblastic Leukemia/Lymphoma in Children/Young Adults
Brief Title: Pilot CAR-T Cells Therapy for Children/Young Adults With CD19+ R/R Leukemia/Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19CAR-T_LL_children
Record Dates: First submitted 2022-04-12; First posted 2022-04-18 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Lymphoblastic B-Cell Lymphoma
Keywords: immunotherapy; CAR-T cells; CD19
MeSH Terms: conditions — Burkitt Lymphoma | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19 CAR-T cells immunotherapy (Experimental): After a cycle of lymphodepleting chemotherapy a patient receive locally produced autologous CD19 CAR-T cells
  Interventions: Biological: CD19 CAR-T-cells; Drug: Tocilizumab

INTERVENTIONS:
Biological: CD19 CAR-T-cells — One dose of CD19 CAR-T cells (1*10e6 CAR+ T-cells/kg) by intravenous infusion.
Drug: Tocilizumab — Before 1h of CAR-T cells infusion a patient receive tocilizumab (8 mg/kg).
  Other Names: Actemra

SUMMARY:
The purpose of this study is to estimate the safety and the efficacy of CAR- T cells immunotherapy for children/young adults with relapsed or refractory acute lymphoblastic leukemia/lymphoma.

DETAILED DESCRIPTION:
Locally manufactured second generation autologous CD19 CAR-T cells are used for immunotherapy. Protocol treatment includes lymphodepleting conditioning (fludarabine + cyclophosphamide) followed by one CAR-T cells intravenous infusion with tocilizumab premedication.

ELIGIBILITY:
Inclusion Criteria:

* CD19+ relapsed or refractory lymphoblastic leukemia/lymphoma;
* Karnofsky or Lansky performance scale greater or equal to 70;
* T-cells count in peripheral blood >150 cells/µL;
* Written informed consent.

Exclusion Criteria:

* primary immunodeficiencies or genetic syndromes;
* neurologic diseases;
* autoimmune diseases or polyallergie;
* transfusion of donor lymphocyte less than 6 week before CAR-T cells infusion;
* GvHD grade 2-4;
* uncontrolled systemic infection;
* hypoxia (Sp02<90%)
* severe hepatic dysfunction: ALT or AST >=3x upper limit of normal for age;
* renal dysfunction: serum creatinine level >=3x upper limit of normal for age;
* positive serology for human immunodeficiency virus (HIV), active hepatite C or B;
* pregnancy.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 month
  Adverse events will be graded according to the CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (CR+CRi+CRm) | 28 days after CAR-T cells infusion
  The proportion of patients with complete remission (CR), CR with incomplete hematologic recovery (CRi), complete molecular remission (CRm).
Overall survival (OS) | 1 year
  The proportion of patients with overall survival
Events free survival (EFS) | 1 year
  Time from CAR-T cells infusion to CR failure, relapse, or death.
Leukemia free survival (LFS) | 1 year
  Time from achievement of CR/CRi/CRm to the time of relapse, death in remission, or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Aleinikova, MD, Prof, Study Director — Belarusian Research Center for Pediatric Oncology, Hematology and Immunology
Locations (1):
- Belarussian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Minsk Oblast, Belarus